CLINICAL TRIAL: NCT00003874
Title: A Phase I/II Study of Combined Enrichment of CD34+ Cells and Depletion of B-Cells From Peripheral Blood Stem Cell Components for Patients With B-Lymphoid Malignancies
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Lymphoma or Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 1345.00; FHCRC-1345.00; NCI-G99-1514; CDR0000067039 (Registry Identifier: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-07-16 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Leukemia; Lymphoma
Keywords: recurrent childhood acute lymphoblastic leukemia; Waldenstrom macroglobulinemia; recurrent childhood lymphoblastic lymphoma; recurrent adult acute lymphoblastic leukemia; refractory chronic lymphocytic leukemia; B-cell chronic lymphocytic leukemia; B-cell childhood acute lymphoblastic leukemia; B-cell adult acute lymphoblastic leukemia; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — ocaratuzumab

INTERVENTIONS:
Biological: monoclonal antibody CD19
Biological: monoclonal antibody CD20
Procedure: in vitro-treated peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Monoclonal antibodies can locate cancer cells and either kill them or deliver cancer-killing substances without harming normal cells.

PURPOSE: Phase I/II trial to study the effectiveness of monoclonal antibody therapy in treating patients who have lymphoma or leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the efficiency of tumor cell removal by immunomagnetic technique in patients with B cell malignancies. II. Determine toxicity of mobilized peripheral blood stem cell (PBSC) components of enriched CD34+ and depleted B cells in this patient population. III. Compare recovery with the use of this treatment regimen to the use of unmanipulated PBSC or CD34+ PBSC components in this patient population.

OUTLINE: Patients are assigned to one of two treatment arms for chemotherapy (chemotherapy protocol following FHCRC-506.2). Patients undergo mobilization and isolation of CD34+ cells as described in FHCRC-506.2. Peripheral blood stem cells are collected by apheresis and the CD34+ cells are isolated using magnetic beads. Monoclonal antibodies to CD19 and CD20 are added to the CD34+ cells to sensitize any remaining tumor cells. Patients undergo transplantation on day 0, according to applicable transplant protocols, one month after mobilization. Some patients may receive posttransplant interleukin-2 after achieving durable engraftment. Patients are followed at day 30, 80, 180, 365, and 395.

PROJECTED ACCRUAL: A total of 20-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed recurrent B cell malignancy that is positive for CD19 and/or CD20 antigens Demonstrated or probable tumor cell contamination of peripheral blood stem cell components No CNS metastases High risk B cell malignancy indicative of autologous hematopoietic stem cell transplantation No HLA matched donors Eligible for mobilization of blood stem cells using chemotherapy and G-CSF Eligible for transplantation on a protocol covering classification and stage of malignancy Intention to proceed to transplantation within 60 days of peripheral blood stem cell collection

PATIENT CHARACTERISTICS: Age: 70 and under Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No active infection HIV negative Adequate organ function as defined in the mobilization and transplant protocols At least 20 CD34+ cells/uL in the peripheral blood before immunomagnetic separation

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-02; Study Completion 2001-09

CONTACTS AND LOCATIONS:
Overall Officials: Scott D. Rowley, MD, FACP, Study Chair — Hackensack University Medical Center Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States